CLINICAL TRIAL: NCT01886820
Title: A Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of [18F]NAV4694 PET for Detection of Cerebral Beta-Amyloid When Compared With Postmortem Histopathology
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Navidea Biopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NAV4-02
Record Dates: First submitted 2013-06-24; First posted 2013-06-26 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Dementia; Alzheimer's Disease
Keywords: Dementia; Alzheimer's Disease; Terminally Ill
MeSH Terms: conditions — Dementia; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [18F]NAV4694 (Experimental): Intravenous [18F]NAV4694 radioactive dose 8.1 mCi(300 MBq) given once
  Interventions: Drug: [18F]NAV4694

INTERVENTIONS:
Drug: [18F]NAV4694

SUMMARY:
To Determine the the Efficacy and Safety of [18F]NAV4694 PET for Detection of Cerebral β-Amyloid When Compared With Postmortem Histopathology

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects will be at least 21 years of age.
* Subjects will have a life expectancy of approximately 6 months
* Subject health is adequate as determined by the investigator to receive [18F]NAV4694
* Female subjects will not be of child-bearing potential or will have a negative urine pregnancy test on day of [18F]NAV4694 injection.
* Must exhibit adequate visual, auditory, and communication capabilities to enable compliance with study procedures. This includes being able to lie down flat in the MRI or CT and PET scanner for a period of approximately 1 hour.
* Subjects must be willing to donate their brains for post mortem examination upon death (this consent can be obtained in the manner specific to the country/region involved).
* Subjects have been fully informed about the study, including provisions of the Health Insurance Portability and Accountability Act (HIPAA), as applicable, and informed consent or assent has been signed and dated (with time) by the subject and/or the subject's legally acceptable representative (LAR) (for individuals with dementia).

Exclusion Criteria:

* Scheduled for surgery and/or another invasive procedure within the time period of up to 7 days after [18F]NAV4694 injection.
* Has severe cerebral macrovascular (i.e., multi-stroke) disease or brain tumor (metastasis/brain cancer) as verified by MRI that prohibits sampling of the required pre-specified ROIs.
* Has any history of any transmissible spongiform encephalopathy (prion disease).
* Has received any contrast material (X-ray, MRI) or radiopharmaceutical within 48 hours prior to, or a therapeutic radiopharmaceutical (e.g., 131-I) within 10 days prior to, or any radiopharmaceutical administration within 10 radioactive half-lives prior to the administration of the investigational product or for whom administration of such substances is planned within 7 days after investigational product administration.
* Is allergic to the investigational product or any of its constituents.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2013-06 (Actual); Primary Completion 2018-06 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of [18F]NAV4694 Brain PET scan positivity compared to histopathology | 6 Months

SECONDARY OUTCOMES:
Quantification of [18F]NAV4694 brain PET Scan positivity compared to histopathology | 6 Months
Incidence of [18F]NAV4694 PET Scan positivity in 6 pre-specified brain regions compared to histopathology | 6 Months
Quantification of [18F]NAV4694 PET Scan positivity in 6 pre-specified brain regions compared to histopathology | 6 Months
Incidence of adverse events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia Reininger, MD PhD, Study Director — Navidea Biopharmaceuticals
Locations (15):
- United States (15):
  - Banner Sun Health Research Institute, Sun City, Arizona
  - University of California San Diego, La Jolla, California
  - Neuropsychiatric Research Center of Southwest Florida, Fort Myers, Florida
  - Mount Sinai Medical Center of Florida, Miami Beach, Florida
  - Galiz Research, Miami Springs, Florida
  - Compass Research, Orlando, Florida
  - Physicians Care Clinical Research, Sarasota, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Biomedical Research Foundation, Shreveport, Louisiana
  - Las Vegas Radiology, Las Vegas, Nevada
  - Albert Einstein College of Medicine, The Bronx, New York
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest Baptist Health-Gerontology, Winston-Salem, North Carolina
  - Valley Medical Center, Centerville, Ohio